CLINICAL TRIAL: NCT03603561
Title: Continuous Theta Burst Transcranial Magnetic Stimulation as an add-on Treatment for Bipolar Depression: a Multicenter Randomized Sham-controlled Trial
Brief Title: Continuous Theta Burst Stimulation as an add-on Treatment for Bipolar Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kaat Hebbrecht, MD, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1808
Record Dates: First submitted 2018-06-05; First posted 2018-07-27 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder; Depression; Mood Disorders; Mental Disorder
Keywords: bipolar depression; TMS; transcranial magnetic stimulation; add-on treatment
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cTBS (Active Comparator)
  Interventions: Device: cTBS
- Sham cTBS (Sham Comparator)
  Interventions: Device: Sham cTBS

INTERVENTIONS:
Device: cTBS — In the cTBS arm, the patients will receive 5 daily session cTBS (5 times uninterrupted train of 900 pulses) separated by a 15 min interval. Patients will be treated with in total 20 cTBS sessions over the right dorsolateral prefrontal cortex, spread over 4 days. A stimulation intensity of 100 % of the resting motor threshold (rMT) of the right abductor pollicis brevis muscle will be used.
  Arms: Active cTBS
Device: Sham cTBS — The sham coil has been specifically developed to mimic the real one but is not associated with a stimulus sensation compared to the coil delivering real stimulation cTBS.
  Arms: Sham cTBS

SUMMARY:
This study aims to investigate the clinical efficacy of continuous theta burst stimulation (cTBS) on the right DLPFC as an add-on treatment in bipolar depression. The study consists of three phases.

Phase 1: Bipolar depressed patients will be selected by a certified psychiatrist, who will administer (semi-)structured clinical interviews (M.I.N.I.-Plus 5.0.0, HRSD-17). The presence of exclusion criteria will be evaluated. Eligible patients will undergo MRI brain imaging for TMS neuronavigation

Phase 2: Baseline clinical, cognitive and psychomotor assessments will take place. Patients will also undergo blood samples for laboratory and research assessments.

TBS involves applying triple-pulse 50 Hz bursts given at a rate of 5 Hz uninterrupted trains (1). Patients will be treated with in total 20 continuous Theta Burst Stimulation (cTBS) session (900 pulses per session) over the right dorsolateral prefrontal cortex, which will be spread over 4 days. A stimulation intensity of 100% of the subject's resting motor threshold (rMT) of the right abductor pollicis brevis muscle will used.

Patients will be randomized to receive either the real cTBS or sham treatment. Sham stimulation will be applied with a sham coil. The sham coil produces identical sounds but is not associated with a stimulus sensation compared to the coil delivering real stimulation cTBS. The investigators expect that real cTBS treatment and not sham will result in a significant and clinical meaningful response.

Phase 3: Two post-treatment assessment moments will take place respectively 3 (max. 4) days and 10 (max. 11) days after the last treatment day. The assessments are the same clinical, cognitive and psychomotor assessments as in phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-IV defined bipolar subjects (bipolar types I and II), depressed or mixed phase, confirmed by the Mini-International Neuropsychiatric Interview (MINI-plus 5.0.0.)
* Hamilton Rating Scale for Depression-17 score of 17 or more.
* Stable psychotropic medication regimen for at least 2 weeks prior to randomization and patient is willing to remain on a stable regimen from screening (S) after the second measurement point T2 (2 to 3 weeks).

Antidepressants:

* On stable antidepressant treatment for 4 weeks.
* Stable antidepressant medication but dose has been recently changed (higher/lower dose): duration of 2 weeks should lie between change of medication dose and screening (S).
* If the patient recently stopped the antidepressant treatment, a wash-out period of 14 days is necessary.

Mood stabilizers:

* On a stable dose of mood-stabilizing medication (e.g., lithium, valproate, carbamazepine, lamotrigine, antipsychotic agents) for at least 4 weeks. In case of change in dose of the mood stabilizing medication, participants can be included given that no or minimal improvement is seen after 2 weeks of dosing.
* Atypical antipsychotics
* On a stable dose of for at least 4 weeks. In case of change in dose of antipsychotics, participants can be included given that no or minimal improvement is seen after 2 weeks of dosing.
* Benzodiazepines are permitted to a maximum allowed dose of equivalent of 40 mg diazepam. If the dosage has been recently changed: stable dose during 2 weeks.
* Able to read, understand and sign the Informed Consent Form.

Exclusion Criteria:

* Contra-indications for TMS treatment:

  * Current or past history of epilepsy.
  * The risk of seizure with any reasons.
  * Organic brain damage (for example mass brain lesions, cerebrovascular accident, …).
  * Neurosurgical interventions.
  * Having a pacemaker or metal or magnetic objects in the brain.
* Unipolar depression
* Psychotic disorder (MINI-plus 5.0.0; DSM-IV codes 295.10, 295.20, .30, .40, .60, .70, .90, 297.10, 298.90); exceptions are: depression with psychotic features MINI-Plus 5.0.0; DSM code 296.23)
* Current alcohol dependence (MINI-plus 5.0.0. DSM IV code 303.9) (in the last year)
* Current substance abuse or dependence (DSM-IV codes 304.00-.90, 305.20 -.70) (in the last year), with the exception of nicotine and caffeine (DSM IV codes 305.10 and 305.90)
* Suicide attempt within 6 months before the start of the study
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in depression severity clinician-rated | Screening, baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Hamilton rating scale for depression (HRSD-17); total scores ranging from 0 to 52. A higher score is indicative of greater depressive pathology

SECONDARY OUTCOMES:
Changes in depression severity self-report | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Beck Depression Inventory (BDI-II); total scores ranging from 0 to 63. Higher total scores indicate more severe depressive symptoms.
Changes in suicidal thoughts - clinician-rated | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Columbia-suicide severity rating scale (total score ranges from 0 to 25; a higher score represent a higher intensity of suicidality)
Changes in cognitive symptoms (1) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Continuous performance test (CPT), a measure of a person's sustained and selective attention: d-prime (the quotient of hits/false alarms that indicate the response sensitivity for discrimination of target from nontarget stimuli). Greater scores represent better ability to distinguish and detect X and non-X stimuli (better sustained attention)
Changes in cognitive symptoms (2) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Symbol Digit Substitution Test (SDST), examining processing speed. Differentiating between the cognitive and the psychomotor processes of slowing (matching time and writing time; msec)
Changes in cognitive symptoms (3) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Stroop test; examining response inhibition (Stroop response interference score)
Changes in psychomotor symptoms (1) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  CORE assessment of psychomotor functioning; total score ranging from 0 to 54. A higher score is indicative of psychomotor impairment (a score of 21 or more is indicative of melancholic depression)
Changes in psychomotor symptoms (2) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Accelometer tool (MotionWatch 8®, CamNtech, Cambridge, UK; measuring gross motor performance): total day activity level (counts per hour). Lower values indicate reduction in gross motor activity. *Cut-off levels from a control group are being collected in another research project of this research group.
Changes in psychomotor symptoms (3) | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Line-copying task (LCT): initiation and movement time (msec)
Change in biological markers (1) | Baseline and 10 days after cTBS or sham (+/- day 14)
  Plasma levels of C reactive protein (CRP)
Change in biological markers (2) | Baseline and 10 days after cTBS or sham (+/- day 14)
  Cytokines (pg/ml)
Change in biological markers (3) | Baseline and 10 days after cTBS or sham (+/- day 14)
  Kynurenines tryptophan catabolites (TRYCAT) levels (mmol/l)
Change in biological markers (4) | Baseline and 10 days after cTBS or sham (+/- day 14)
  Brain-derived neurotrophic factor (BDNF; ng/ml)
Differences in adverse events following cTBS or sham - self report | 3 days after cTBS or sham (+/- day 7)
  Adverse effects questionnaire
Differences in development of (hypo)manic symptoms | Baseline, 3 days after cTBS or sham (+/- day 7), 10 days after cTBS or sham (+/- day 14)
  Young mania rating scale (YMRS): evaluates the presence and severity of mania. The score ranges from 0 to 60. Scores higher than 12 are indicative for mania, scores of 2 or lower indicate euthymia.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospital of Brussels, Brussels
  - University Psychiatric Hospital Duffel, Duffel

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172